CLINICAL TRIAL: NCT02807727
Title: Randomised Control Study on Cardiac Protection With Intralipid® in Patients Undergoing Coronary Artery Bypass Grafting on Cardiopulmonary Bypass
Brief Title: Cardiac REperfusion With Intralipid® at Reperfusion
Acronym: CREW-I
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nkanyiso Hadebe (Other)
Responsible Party: Sponsor-Investigator, Nkanyiso Hadebe, Dr, University of Cape Town
Organization: University of Cape Town (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CREW-I
Record Dates: First submitted 2016-06-13; First posted 2016-06-21 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intralipid 20% (Active Comparator): Intravenous single bolus of 1.5 ml/kg of Intralipid 20% over 3 minutes.
  Interventions: Drug: Intralipid 20%
- Modified Ringers Lactate (Placebo Comparator): Intravenous single bolus of 1.5 ml/kg of MRL over 3 minutes.
  Interventions: Drug: Modified Ringers Lactate

INTERVENTIONS:
Drug: Intralipid 20% — Single intravenous bolus dose of 1.5 ml/kg over 3 minutes
  Other Names: Lipid Emulsion 20%
  Arms: Intralipid 20%
Drug: Modified Ringers Lactate — Single intravenous bolus dose of 1.5 ml/kg over 3 minutes
  Other Names: MRL
  Arms: Modified Ringers Lactate

SUMMARY:
This study will evaluate the benefit of Intralipid® or placebo administered prior to reperfusion to limit ischemia reperfusion injury as measured by the geometric mean difference of the release of troponin I over 72 hours after coronary artery bypass.

DETAILED DESCRIPTION:
A single center randomised control study on cardiac protection with INTRALIPD in patients undergoing coronary artery bypass grafting on cardiopulmonary bypass.

Purpose and objectives:

Reperfusion after coronary artery bypass grafting is associated with a modifiable leak in cardiac Troponin I (cTnI) secondary to ischemia reperfusion injury. The purpose of the study is to test whether INTRALIPID administered at reperfusion can limit myocardial reperfusion injury as measured by cTnI release in patients undergoing coronary artery bypass grafting.

Trial design:

This study is a prospective single centre double blind placebo controlled randomised trial.

Sample size: 30 Adult Male and Female Patients

Investigational drug(s):

INTRALIPID 20% Fresenius Kabi (SA) Registration Number: K/25.2/316 Formulation: IV Solution Strength: 20% (200mg/ml) Modified Ringer's Lactate Fresenius Kabi (SA) Registration Number: C/24/218 Formulation: IV Solution Dose for both drugs: 1.5 ml/kg Administration: IV Bolus through CVP Blood sampling and tissue biopsies: cTnI will be sampled at fixed time points, baseline 1, 6, 9, 12, 24, 48, and 72 hours after surgery. The first biopsy will be done prior to cardioplegic arrest and the second biopsy will be done 5 minutes after reperfusion.

Safety assessments:

The safety of the interventions will be monitored routinely for all patients and these will focus on:

1. Changes in the lipid profile after Intralipid
2. Coagulation as measured by ACT, TEG and PFA
3. Oxygenation with Arterial Blood Gas monitoring
4. Hemodynamic monitoring and echocardiography
5. Lipid interference with laboratory measurements. The laboratory will be informed on specimen preparation to avoid interference with instruments
6. Post operative hemodynamic Intensive Care Unit Monitoring Measurement will be reported on all safety monitoring and will be considered adverse events where the measured parameter results are out of range from the laboratory references.

Efficacy assessments. Primary endpoint: The efficacy of the drug will be determined by the geometric mean (95% CI) difference in the AUC of the cTnI concentration calculated according to the trapezoid rule.

Secondary End Point: Exploring the molecular mechanism involved in cardiac protection by analyzing tissue sample differences in the phosphorylation cytoplasmic protein kinase.

ELIGIBILITY:
Inclusion Criteria:

* First time elective isolated CABG
* Ejection Fraction greater the 40 by echocardiography or subjectively judged as preserved or good by ventriculography.
* Male and female adults between 18 and 65 years of age.
* Women must have a negative serum pregnancy test at screening.
* Body mass Index (BMI) between 21 and 35 kg/m2.
* Baseline clinical laboratory tests at screening within the reference ranges

Exclusion Criteria:

* Received an investigational drug or participated in another research trial within 30 days before the first dose of trial drug or at any time throughout the trial.

  * Evidence of current or history of clinically significant oncologic, pulmonary, hepatic with elevated liver functions enzymes 1.5* Upper Limit of Normal (ULN), cardiovascular, haematologic, metabolic, neurological, immunologic, nephrologic, endocrine particularly Diabetes Mellitus as defined by the American Diabetic Association, psychiatric disease, or clinically significant current infection.
  * Patients with renal impairment with a creatinine greater than 200 μmol/L
  * Evidence of current or history of clinically significant gastrointestinal (excluding appendectomy, cholecystectomy) disease.
  * Myocardial infarction within the previous 2 weeks.
  * Patients who require inotropic or mechanical cardiac support prior to anaesthesia.
  * Contraindication to the trial drugs Previous Hypertriglyceridemia pancreatitis. Hypertriglyceridemia with plasma triglyceride levels > 5.7mmol/L Egg, peanut and soybean allergy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of the serum Troponin I Leak over 72 hours | Over 72 hours
  The primary endpoint will be assessed by the geometric mean (95% CI) difference between the protocol and control groups of the area under the curve for the cTnI concentration in serum over 72 hours (sampled at 1, 6, 12, 24, 48 and 72 hours) calculated according to the trapezoid rule.

SECONDARY OUTCOMES:
Signaling Pathways of intralipid induced cardiac protection | 5 minutes after reperfusion
  Two right atrial and two left ventricular biopsies will be collected before cardioplegia and the second will be collected 5 minutes prior to reperfusion. These will be used to compare the activation of signalling protein between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nkanyiso E Hadebe, MBBCh, Study Chair — University of Cape
Locations (1):
- Department of Anaesthesia, Groote Schuur Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared

REFERENCES:
- [Derived] Hadebe N, Cour M, Imamdin A, Petersen T, Pennel T, Scherman J, Snowball J, Ntsekhe M, Zilla P, Swanevelder J, Lecour S. Cardioprotection with Intralipid During Coronary Artery Bypass Grafting Surgery on Cardiopulmonary Bypass: A Randomized Clinical Trial. Cardiovasc Drugs Ther. 2025 Oct;39(5):1045-1052. doi: 10.1007/s10557-024-07594-w. Epub 2024 Jun 12. PMID 38864969